CLINICAL TRIAL: NCT06927024
Title: A Randomized, Sham-controlled Pilot Trial of a Novel Therapeutic Strategy (taVNS) for Autonomic Nervous System (ANS) Dysfunction in Chronic Kidney Disease (CKD)
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) in Chronic Kidney Disease (CKD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-00756; 1K23DK139462-01A1 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Experimental): Participants receive two weeks of 15-minute taVNS daily in the morning.
  Interventions: Device: Active taVNS
- Sham taVNS (Sham Comparator): Participants receive two weeks of 15-minute sham intervention daily in the morning.
  Interventions: Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — Active taVNS delivered via the TENS Device 7000.
  Arms: Active taVNS
Device: Sham taVNS — Sham taVNS delivered via the TENS Device 7000.
  Arms: Sham taVNS

SUMMARY:
30 patients will participate in a prospective randomized clinical trial to test the safety, tolerability and efficacy of transcutaneous auricular vagus nerve stimulation (taVNS) for autonomic nervous system (ANS) dysfunction in the chronic kidney disease (CKD) stage 3-5 setting.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age ≥18 years
* Diagnosis of Chronic Kidney Disease (CKD) stage 3-5 [estimated glomerular filtration rate &le;60 mL/min/1.73m2]
* Receiving care at NYU Nephrology outpatient practice
* Able to provide informed consent

Exclusion Criteria:

* Primary ANS disorders (e.g., Parkinson's disease)
* Arrhythmias
* Implantable cardioverter-defibrillator (ICD) or pacemaker (PPM) precluding assessment of HRV (e.g., chronic atrial fibrillation)
* On maintenance dialysis (HD)
* Epilepsy
* Symptomatic bradycardia
* Presence of an implantable defibrillators
* Presence of a permanent pacemaker
* Unable to consent
* Incarcerated individuals
* Pregnant individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients who Complete 2 Weeks of Intervention | Week 2
  Proportion of patients who use the device for 2 weeks (14 sessions). Measure of feasibility.
Proportion of Patients who Tolerate Each Full 15-Minute Session | Week 2
  Proportion of patients who use the device for 2 weeks (14 sessions), 15 minutes per session. Measure of feasibility
Incidence of Severe Bradycardia following taVNS Use | Up to Week 2
  Severe bradycardia defined as heart rate (HR) <50 beats per minute. Measure of safety.
Incidence of Severe Tachycardia following taVNS Use | Up to Week 2
  Severe tachycardia defined as heart rate (HR) >100 beats per minute. Measure of safety.
Incidence of Syncope following taVNS Use | Up to Week 2
  Measure of safety.

SECONDARY OUTCOMES:
Proportion of eligible patients who consent to use the device for 2 weeks | Up to Week 2
  Also known as "recruitment yield." Measure of feasibility.
Change in High Frequency (HF) Signal from Baseline | Baseline, Week 2
  HF defined as vagal heart rate variation (HRV) modulation. Measure of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Qandeel Soomro, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Qandeel.Soomro@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Qandeel.Soomro@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.